CLINICAL TRIAL: NCT00253916
Title: Exercise in Men Receiving Radiation Therapy for Prostate Cancer: Effects on Fatigue, Toxicity, Body Composition, Muscular Fitness, Cardiorespiratory Fitness and Quality of Life.
Brief Title: Exercise in Men Receiving Radiation Therapy for Prostate Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Cancer Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCIC 013232; OTT 02-04 (Other: OHRI); CERHO 2002263-01H (Other: OHRI)
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (3):
- Control Arm (No Intervention): No exercise measured
- Aerobic cardiovascular exercise program (Experimental): Aerobic cardiovascular exercise program
  Interventions: Behavioral: Aerobic cardiovascular exercise program
- Resistance Exercise Program (Experimental): Resistance Exercise Program
  Interventions: Behavioral: Resistance Exercise Program

INTERVENTIONS:
Behavioral: Aerobic cardiovascular exercise program — Aerobic cardiovascular exercise program
  Arms: Aerobic cardiovascular exercise program
Behavioral: Resistance Exercise Program — Resistance Exercise Program
  Arms: Resistance Exercise Program

SUMMARY:
Androgen Deprivation Therapy is a commonly used treatment for men with Prostate Cancer. Unfortunately this can lead to functional decline, fatigue, increased body fatness, loss of lean body tissue and impaired QOL. Previous research has demonstrated the exercise can may reduce fatigue and improve QOL in men on ADT. This study will evaluate whether aerobic versus resistance exercise over a 24 week period of training will reduce morbidity and improve QOL in men receiving radiation plus or minus ADT with curative intent

DETAILED DESCRIPTION:
A total of 220 men with a diagnosis of prostate cancer, scheduled to receive radiation will be recruited. The study is a parallel 3-group design with groups stratified for intended duration of ADT ( greater or less than 12 weeks) and random assignment to aerobic, resistance or Wait List control groups. The dependent variable of interest will fatigue measured at 24 weeks by the 13 item FACT-Fatigue. Dependent variables of secondary interest will be toxicity of radiation, body composition, muscular fitness, cardio-respiratory fitness, metabolic fitness, and prostate specific QOL. All exercise sessions will be performed 3 times per week at the Ottawa Hospital regional Cancer Center

ELIGIBILITY:
Inclusion Criteria:

* Prostate Cancer
* Radiation Therapy with curative Intent
* ADT

Exclusion Criteria:

* Contraindication to exercise
* Uncontrolled hypertension
* Uncontrolled Cardiac Disease
* Uncontrolled psychotic condition
* Unable to obtain informed consent

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2002-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Fatigue- FACT F | 24 weeks

SECONDARY OUTCOMES:
Toxicity of Radiotherapy Body Composition Muscular Fitness Cardiorespiratory Fitness Metabolic Fitness Prostate Specific QOL | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roanne Segal, Principal Investigator — OHRI
Locations (1):
- The Ottawa Hospital-Integrated Cancer Program, Ottawa, Ontario, Canada

REFERENCES:
- [Result] Segal RJ, Reid RD, Courneya KS, Malone SC, Parliament MB, Scott CG, Venner PM, Quinney HA, Jones LW, D'Angelo ME, Wells GA. Resistance exercise in men receiving androgen deprivation therapy for prostate cancer. J Clin Oncol. 2003 May 1;21(9):1653-9. doi: 10.1200/JCO.2003.09.534. PMID 12721238